CLINICAL TRIAL: NCT02411578
Title: Mini-Dose Glucagon for Adults With Type 1 Diabetes: A Study to Assess the Efficacy and Safety of Mini-dose Glucagon for Treatment of Non-severe Hypoglycemia in Adults With Type 1 Diabetes
Brief Title: Mini-Dose Glucagon to Treat Non-Severe Hypoglycemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: T1DX Mini-dose Non-Severe
Record Dates: First submitted 2015-03-27; First posted 2015-04-08 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; Type 1 diabetes; Mini-dose glucagon; adults; non-severe hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-Pen Mini™ (glucagon injection) (Experimental): Participants are to check blood glucose (BG) with study meter once their continuous glucose monitor (CGM) reads <70 mg/dl or they experience symptoms. Participants will be instructed to treat using mini-dose glucagon for certain phases/periods when BG is 40 to 69 mg/dl (considered a non-severe hypoglycemic event).
  For every event, participant will check BG with meter 3 times and treat according to protocol instructions based on BG measurement.
  Interventions: Drug: G-Pen Mini™ (glucagon injection)
- Glucose Tabs (Active Comparator): Participants are to check their blood glucose (BG) with study meter once their continuous glucose meter reads <70 mg/dl or they experience symptoms. Participants will be instructed to treat using oral glucose tablets for certain phases/periods when BG is 40 to 69 mg/dl (considered a non-severe hypoglycemic event).
  For every event, participant will check BG with meter 3 times and treat according to protocol instructions based on BG measurement.
  Interventions: Other: Glucose Tablets

INTERVENTIONS:
Drug: G-Pen Mini™ (glucagon injection) — 1st BG check, 1st treatment
  1. BG is 50-69 mg/dl, treatment is 150 µg of glucagon
  2. BG is 40-49 mg/dl, treatment is 300 µg of glucagon
  15 min later, 2nd BG check, 2nd treatment
  1. BG is 60-69 mg/dl, no treatment
  2. BG is 50-59 mg/dl, treatment is 150 µg of glucagon
  3. BG is <50 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  30 minutes later, 3rd BG check, 3rd treatment
  1. BG is >=70, no treatment
  2. BG is <70 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  (150 µg of glucagon per syringe)
  Other Names: mini-dose glucagon
  Arms: G-Pen Mini™ (glucagon injection)
Other: Glucose Tablets — 1st BG check, 1st treatment
  1. BG is 50-69 mg/dl, treatment is 15 grams of carbohydrates
  2. BG is 40-49 mg/dl, treatment is 30 grams of carbohydrates
  15 min later, 2nd BG check, 2nd treatment
  1. BG is 60-69 mg/dl, no treatment
  2. BG is 50-59 mg/dl, treatment is 15 grams of carbohydrates
  3. BG is <50 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  30 minutes later, 3rd BG check, 3rd treatment
  1. BG is >=70, no treatment
  2. BG is <70 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  (5 grams of fast-acting carbohydrates (D-Glucose) per tablet)
  Other Names: over-the-counter oral glucose tablets; glucose tabs
  Arms: Glucose Tabs

SUMMARY:
The purpose of this study is to determine if a small dose of glucagon (mini-dose glucagon) is effective for the treatment of non-severe hypoglycemia in adults with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
There are three phases included in this study: (1) Pre-crossover Trial Run-in Phase, (2) Randomized Clinical Trial (RCT) Crossover Trial Phase, and (3) Post-Crossover Trial Extension Phase.

1. Run-in Phase:

   Prior to commencing the crossover trial, study enrollment will begin with a 2 week run-in phase to assess hypoglycemia eligibility and compliance.
2. Crossover Trial Phase:

   The Crossover Trial Phase will consist of two (3-week) periods.

   The Crossover Trial Phase will include up to 24 participants who complete these study periods. Participants who do not complete both periods or who do not have at least one event during both periods may be replaced.

   During the Crossover Trial Phase participants will be randomized into two groups: (1) Group A will use mini-dose glucagon in period 1 and oral glucose tablets in period 2 and (2) Group B will use oral glucose tablets in period 1 and mini-dose glucagon in period 2. Each group with follow the applicable treatment arm according to their randomized group.
3. Extension Phase:

The Post-Crossover Trial phase will commence upon completion of the second 3-week period of the Crossover Trial Phase. Participants will have a 3 week phase during which time they will decide whether to use mini-dose glucagon or glucose tablets to treat each non-severe hypoglycemic event or to prevent hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of presumed autoimmune T1D and receiving daily insulin
2. Age: 18.0 to < 65.0 years
3. Duration of T1D: ≥2.0 years
4. Body mass index 20.0 to <35.0 kg/m2 and weight 110 to <250 lbs
5. HbA1c <8.5% (point of care or local lab, within past month)
6. Using continuous subcutaneous insulin infusion (CSII) therapy (i.e., insulin pump) for at least 3 months, with no plans to discontinue use during the study (and no use of active low glucose suspend feature within the last 4 weeks)
7. Using continuous glucose monitor ≥6 days/week in the last 4 weeks, with no plans to discontinue continuous glucose monitor use during the study
8. Continuous glucose monitor glucose level <70 mg/dl during daytime hours (e.g., 8am - 10pm) on at least 7 of the past 28 days (a modification can be made for participants with non-traditional waking hours) evaluated from downloaded CGM data
9. Females must meet one of the following criteria:

   * Of childbearing potential and not currently pregnant (negative pregnancy test) or lactating, and agrees to use an accepted contraceptive regimen as described in the study procedure manual throughout the entire duration of the study (from screening visit until study completion); or
   * Of non-childbearing potential, defined as a female who has had a hysterectomy or tubal ligation, is clinically considered infertile or is in a menopausal state (at least 1 year without menses)
10. In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
11. Willing to adhere to the protocol requirements for the duration of the study
12. Participant has a smart phone available and is able to use it daily
13. Must be enrolled in the T1D Exchange clinic registry or willing to join the clinic registry

Exclusion Criteria:

1. More than 1 severe hypoglycemic episode in the past 12 months (as defined by an episode that required third party assistance for treatment)
2. More than 1 episode of diabetic ketoacidosis in the past 12 months (as defined by an episode diagnosed as diabetic ketoacidosis that required treatment in an emergency department or hospitalization)
3. Presence of cardiovascular, gastrointestinal, liver or kidney disease, or any medical condition which, in the judgment of the investigator, could potentiate or predispose to undesired effects or could interfere with the absorption, distribution, metabolism, or excretion of glucagon or ability to respond appropriately to mild to moderate hypoglycemia.
4. Known presence of hereditary problems of glycogen storage disease, galactose and/or lactose intolerance
5. Males with alcohol use in excess of 3 or more drinks per day, on average and females with alcohol use in excess of 2 or more drinks per day, on average
6. Use of non-insulin anti-diabetic medications
7. Use of daily systemic beta-blocker
8. Use of beta-adrenergic agonists, theophylline (or other methylxanthines)
9. Use of 1st generation anticholinergic drugs (such as Brompheniramine, Chlorpheniramine, Dimenhydrinate, Diphenhydramine, and Doxylamine)
10. Use of systemic corticosteroids
11. History of hypersensitivity to glucagon or any related product or excipient or severe hypersensitivity reactions (such as angioedema) to any drugs
12. History of epilepsy or seizure disorder
13. Uncontrolled hypertension, >160 mmHg systolic or >100 mmHg diastolic
14. Currently a high endurance exerciser or plans to perform high endurance exercise during study (from screening visit until study completion)

    * High endurance exerciser defined as a person who regularly competes in running, cycling, rowing, swimming or any other endurance-based activity for the purpose of competition (>2100 metabolic equivalent of task (MET) minutes per week [i.e. 7 METs x 60 minutes x 5 days a week, where 7 METs is equivalent to jogging])
15. Currently following a very low calorie or other weight-loss diet
16. Participation in other studies involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before screening for the current study or planning to participate in another such study during participation in the current study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morey W Haymond, MD, Study Chair — Baylor College of Medicine; Stephanie N DuBose, MPH, Principal Investigator — Jaeb Center for Health Research
Locations (5):
- United States (5):
  - University of Colorado/Barbara Davis Center for Diabetes, Aurora, Colorado
  - Yale University of Medicine, New Haven, Connecticut
  - Joslin Diabetes Center, Boston, Massachusetts
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Cryer PE. The barrier of hypoglycemia in diabetes. Diabetes. 2008 Dec;57(12):3169-76. doi: 10.2337/db08-1084. No abstract available. PMID 19033403
- [Background] Cryer PE. Hypoglycemia in type 1 diabetes mellitus. Endocrinol Metab Clin North Am. 2010 Sep;39(3):641-54. doi: 10.1016/j.ecl.2010.05.003. PMID 20723825
- [Background] Raju B, Arbelaez AM, Breckenridge SM, Cryer PE. Nocturnal hypoglycemia in type 1 diabetes: an assessment of preventive bedtime treatments. J Clin Endocrinol Metab. 2006 Jun;91(6):2087-92. doi: 10.1210/jc.2005-2798. Epub 2006 Feb 21. PMID 16492699
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Beck RW, Hirsch IB, Laffel L, Tamborlane WV, Bode BW, Buckingham B, Chase P, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Huang ES, Kollman C, Kowalski AJ, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer SA, Wilson DM, Wolpert H, Wysocki T, Xing D. The effect of continuous glucose monitoring in well-controlled type 1 diabetes. Diabetes Care. 2009 Aug;32(8):1378-83. doi: 10.2337/dc09-0108. Epub 2009 May 8. PMID 19429875
- [Background] Haymond MW, Schreiner B. Mini-dose glucagon rescue for hypoglycemia in children with type 1 diabetes. Diabetes Care. 2001 Apr;24(4):643-5. doi: 10.2337/diacare.24.4.643. PMID 11315823
- [Background] Hartley M, Thomsett MJ, Cotterill AM. Mini-dose glucagon rescue for mild hypoglycaemia in children with type 1 diabetes: the Brisbane experience. J Paediatr Child Health. 2006 Mar;42(3):108-11. doi: 10.1111/j.1440-1754.2006.00807.x. PMID 16509909
- [Background] Hasan KS, Kabbani M. Mini-dose glucagon is effective at diabetes camp. J Pediatr. 2004 Jun;144(6):834. No abstract available. PMID 15212060
- [Derived] Haymond MW, DuBose SN, Rickels MR, Wolpert H, Shah VN, Sherr JL, Weinstock RS, Agarwal S, Verdejo AS, Cummins MJ, Newswanger B, Beck RW; T1D Exchange Mini-dose Glucagon Study Group. Efficacy and Safety of Mini-Dose Glucagon for Treatment of Nonsevere Hypoglycemia in Adults With Type 1 Diabetes. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2994-3001. doi: 10.1210/jc.2017-00591. PMID 28591776
- See also: Safety and Efficacy Study of Mini-Dose Glucagon (G-Pen Mini) in Patients With Type 1 Diabetes — https://clinicaltrials.gov/ct2/show/NCT02081014?term=Xeris+G-Pen&rank=1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 consented for Run-in; 1 ineligible after consent; 2 ineligible after Run-in phase; 3 withdrew
Groups:
- G-Pen Mini™ (Glucagon Injection), Then Glucose Tabs: For G-Pen Mini Period:
  Participants are to check blood glucose (BG) with study meter if continuous glucose monitor (CGM) reads <70 mg/dl or they experience symptoms. Participants instructed to treat using mini-dose glucagon for certain phases/periods when BG is 40 to 69 mg/dl (considered a non-severe hypoglycemic event).
  G-Pen Mini™ (glucagon injection): 1st BG check, 1st treatment
  1. BG is 50-69 mg/dl, treatment is 150 µg of glucagon
  2. BG is 40-49 mg/dl, treatment is 300 µg of glucagon
  15 min later, 2nd BG check, 2nd treatment
  1. BG is 60-69 mg/dl, no treatment
  2. BG is 50-59 mg/dl, treatment is 150 µg of glucagon
  3. BG is <50 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  30 minutes later, 3rd BG check, 3rd treatment
  1. BG is >=70, no treatment
  2. BG is <70 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
- Glucose Tabs, Then G-Pen Mini: For Glucose Tabs Period:
  Participants are to check blood glucose (BG) with study meter if continuous glucose meter reads <70 mg/dl or they experience symptoms. Participants instructed to treat using oral glucose tablets for certain phases/periods when BG is 40 to 69 mg/dl (considered a non-severe hypoglycemic event).
  Glucose Tabs: 1st BG check, 1st treatment:
  1. BG is 50-69 mg/dl, treatment is 15 grams of carbohydrates
  2. BG is 40-49 mg/dl, treatment is 30 grams of carbohydrates
  15 min later, 2nd BG check, 2nd treatment
  1. BG is 60-69 mg/dl, no treatment
  2. BG is 50-59 mg/dl, treatment is 15 grams of carbohydrates
  3. BG is <50 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  30 minutes later, 3rd BG check, 3rd treatment
  1. BG is >=70 mg/dl, no treatment
  2. BG is <70 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
Period: Crossover Trial Phase
Arm/Group | G-Pen Mini™ (Glucagon Injection), Then Glucose Tabs | Glucose Tabs, Then G-Pen Mini
Started | 8 | 12
Completed | 8 | 11
Not Completed | 0 | 1
Not completed — Pregnancy | 0 | 1
Period: Extension Phase
Arm/Group | G-Pen Mini™ (Glucagon Injection), Then Glucose Tabs | Glucose Tabs, Then G-Pen Mini
Started | 8 | 9 (2 Crossover Trial participants could not continue due to study syringes expiration)
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Characteristics of the 16 participants with analyzable hypoglycemic events (1 of 20 participants randomized was dropped due to pregnancy and 3 participants did not have any analyzable hypoglycemic events.)
Groups:
- Total: Total of all reporting groups
Arm/Group | G-Pen Mini™ (Glucagon Injection), Then Glucose Tabs | Glucose Tabs, Then G-Pen Mini | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (9.1) | 36.9 (12.2) | 38.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 10 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 6.9 (0.6) | 7.4 (0.9) | 7.2 (0.8)
Duration of Type 1 Diabetes [Mean (Standard Deviation); unit: years] | 24.8 (14.2) | 22.5 (15.8) | 23.4 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Hypoglycemic Events ≥50 mg/dl 15 Minutes AND ≥ 70 mg/dl 30 Minutes After Initial Treatment
Time Frame: 30 minutes
Population: Limited to events with starting BG of 50-69 mg/dL
Measure: Count of Units; unit: Hypoglycemic Events
Units Other Than Participants: Hypoglycemic Events
Groups:
- G-Pen Mini™ (Glucagon Injection): For G-Pen Mini period:
  Participants are to check blood glucose (BG) with study meter if continuous glucose monitor (CGM) reads <70 mg/dl or they experience symptoms. Participants instructed to treat using mini-dose glucagon for certain phases/periods when BG is 40 to 69 mg/dl (considered a non-severe hypoglycemic event).
  G-Pen Mini™ (glucagon injection): 1st BG check, 1st treatment
  1. BG is 50-69 mg/dl, treatment is 150 µg of glucagon
  2. BG is 40-49 mg/dl, treatment is 300 µg of glucagon
  15 min later, 2nd BG check, 2nd treatment
  1. BG is 60-69 mg/dl, no treatment
  2. BG is 50-59 mg/dl, treatment is 150 µg of glucagon
  3. BG is <50 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  30 minutes later, 3rd BG check, 3rd treatment
  1. BG is >=70, no treatment
  2. BG is <70 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
- Glucose Tabs: For Glucose Tabs Period:
  Participants are to check blood glucose (BG) with study meter if continuous glucose meter reads <70 mg/dl or they experience symptoms. Participants instructed to treat using oral glucose tablets for certain phases/periods when BG is 40 to 69 mg/dl (considered a non-severe hypoglycemic event).
  Glucose Tabs: 1st BG check, 1st treatment:
  1. BG is 50-69 mg/dl, treatment is 15 grams of carbohydrates
  2. BG is 40-49 mg/dl, treatment is 30 grams of carbohydrates
  15 min later, 2nd BG check, 2nd treatment
  1. BG is 60-69 mg/dl, no treatment
  2. BG is 50-59 mg/dl, treatment is 15 grams of carbohydrates
  3. BG is <50 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  30 minutes later, 3rd BG check, 3rd treatment
  1. BG is >=70 mg/dl, no treatment
  2. BG is <70 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 16 | 16
Number analyzed (Hypoglycemic Events) | 62 | 56
Hypoglycemic Events | 58 | 53
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; For the crossover trial primary analysis, analyzed events were study treatment events meeting the following criteria: a) a survey was completed in the smart phone application, b) the initial BG measurement was 40 to 69 mg/dL, c) BG measurements were performed at both the 15-minute (in a window of 13 to 20 minutes) and 30-minute (28 to 40 minutes) time points, and d) appropriate treatment including dose was taken both at the initial and 15-minute time points; Test type: Superiority; p = 0.99, Mixed Models Analysis — Proportions of successes in each arm were compared using a generalized linear mixed model with a logistic link function, random participant effect to account for correlated data from some pts having multiple events, and adjustment for baseline BG

2. Secondary Outcome: Continuous Glucose Monitor (CGM) Minimum Glucose, Event Level
Description: Minimum glucose from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first hour after start of hypoglycemic event
Time Frame: 60 Minutes
Population: A participant had to have sufficient calibrations using study BGM to compare BGM and CGM data to ensure matching dates and times. Event level requirements: 1) initial treatment and dose had to be correct, 2) ≥6 CGM readings within 1 hour after initial treatment, and 3) first CGM glucose after the start of the hypoglycemic event had to be <80 mg/dL
Measure: Median (Inter-Quartile Range); unit: mg/dL
Units Other Than Participants: Hypoglycemic Events
Groups:
- G-Pen Mini™ (Glucagon Injection): For G-Pen Mini Period:
  Participants are to check blood glucose (BG) with study BG meter (BGM) if continuous glucose monitor (CGM) reads <70 mg/dl or they experience symptoms. Participants instructed to treat using mini-dose glucagon for certain phases/periods when BG is 40 to 69 mg/dl (considered a non-severe hypoglycemic event).
  G-Pen Mini™ (glucagon injection): 1st BG check, 1st treatment
  1. BG is 50-69 mg/dl, treatment is 150 µg of glucagon
  2. BG is 40-49 mg/dl, treatment is 300 µg of glucagon
  15 min later, 2nd BG check, 2nd treatment
  1. BG is 60-69 mg/dl, no treatment
  2. BG is 50-59 mg/dl, treatment is 150 µg of glucagon
  3. BG is <50 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
  30 minutes later, 3rd BG check, 3rd treatment
  1. BG is >=70, no treatment
  2. BG is <70 mg/dl, treatment is participant's preferred oral carbohydrate and not mini-dose glucagon
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
mg/dL | 59 [52 to 66] | 56 [52 to 60]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.34, Mixed Models Analysis; Analyzed with generalized linear mixed model with an identity link. Due to violations of normality, rank transformations were used in model

3. Secondary Outcome: CGM Maximum Glucose, Event Level
Description: Maximum glucose from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first hour after start of hypoglycemic event
Time Frame: 60 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
mg/dL | 102 [83 to 119] | 116 [98 to 143]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.01, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: CGM Mean Glucose, Event Level
Description: Median (IQR) reported for mean glucose from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first hour after start of hypoglycemic event
Time Frame: 60 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
mg/dL | 79 [69 to 91] | 87 [77 to 102]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.02, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: CGM Time in Range, Event Level
Description: Percentage of time 70-180 mg/dL from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first hour after start of hypoglycemic event
Time Frame: 60 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
percentage of time | 62 [42 to 79] | 67 [58 to 71]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.86, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: CGM Time Below 70 mg/dL, Event Level
Description: Percentage of time <70 mg/dL from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first hour after start of hypoglycemic event
Time Frame: 60 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
percentage of time | 35 [13 to 58] | 33 [26 to 42]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.95, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: CGM Minimum Glucose, Event Level
Description: Minimum glucose from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first 2 hours after start of hypoglycemic event
Time Frame: 120 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
mg/dL | 57 [51 to 65] | 56 [52 to 60]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.78, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

8. Secondary Outcome: CGM Maximum Glucose, Event Level
Description: Maximum glucose from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first 2 hours after start of hypoglycemic event
Time Frame: 120 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
mg/dL | 122 [102 to 159] | 139 [116 to 161]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.21, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

9. Secondary Outcome: CGM Mean Glucose, Event Level
Description: Median (IQR) reported for mean glucose from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first 2 hours after start of hypoglycemic event
Time Frame: 120 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
mg/dL | 95 [77 to 113] | 108 [89 to 119]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.09, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

10. Secondary Outcome: CGM Time in Range, Event Level
Description: Percentage of time 70-180 mg/dL from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first 2 hours after start of hypoglycemic event
Time Frame: 120 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
percentage of time | 79 [50 to 88] | 79 [69 to 86]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.49, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

11. Secondary Outcome: CGM Time Below 70 mg/dL
Description: Percentage of time <70 mg/dL from CGM data, following each hypoglycemic event with starting BG 50-69 mg/dL, during first 2 hours after start of hypoglycemic event
Time Frame: 120 Minutes
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
Number analyzed (Hypoglycemic Events) | 48 | 36
percentage of time | 20 [9 to 40] | 19 [13 to 25]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.63, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

12. Secondary Outcome: CGM Mean Glucose
Description: Median (IQR) reported for mean glucose from CGM data computed over entire 3 weeks of treatment period
Time Frame: 3 weeks
Population: Limited to participants who had at least 72 hours of CGM data during each period
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
mg/dL | 143 [135 to 169] | 149 [136 to 177]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.41, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

13. Secondary Outcome: CGM Time in Range
Description: Percentage of time 70-180 mg/dL from CGM data computed over entire 3 weeks of treatment period
Time Frame: 3 weeks
Population: Limited to participants who had at least 72 hours of CGM data during each period
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
percentage of time | 71 [60 to 79] | 71 [57 to 79]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.80, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

14. Secondary Outcome: CGM Time Below 70
Description: Percentage of time <70 mg/dL from CGM data computed over entire 3 weeks of treatment period
Time Frame: 3 weeks
Population: Limited to participants who had at least 72 hours of CGM data during each period
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
percentage of time | 5 [2 to 7] | 4 [2 to 6]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.13, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

15. Secondary Outcome: CGM Coefficient of Variation
Description: Coefficient of Variation from CGM data computed over entire 3 weeks of treatment period
Time Frame: 3 weeks
Population: Limited to participants who had at least 72 hours of CGM data during each period
Measure: Median (Inter-Quartile Range); unit: percentage coefficient of variation
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 15 | 15
percentage coefficient of variation | 35 [33 to 40] | 36 [35 to 39]
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.70, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

16. Post Hoc Outcome: Clinical Grading - Limited to Events in Primary Analysis
Description: 2 graders, blinded to treatment arm, independently graded each hypoglycemic event as a clinical failure or success based on all available BG concentrations within 1 hour of initial treatment. All BG values, along with corresponding time elapsed since treatment, were reviewed to determine whether the response would be considered a treatment success, in a clinical setting. There were no specific cut points; rather than basing the success criteria on whether the BG was above specific cutpoints by specific times, the grader decided whether the event would be considered a success in a clinical setting (i.e. if the BG increased after treatment and reached and maintained a satisfactory level after the treatment). The graders to achieve a consensus grading adjudicated discordant gradings (6% of events). The number of events graded as a treatment success were reported out of the total number of hypoglycemic events, for each treatment arm.
Time Frame: 60 minutes
Population: Analysis was limited to hypoglycemic events included in the primary analysis. 3 hypoglycemic events were deemed Indeterminate by the graders during the glucagon period.
Measure: Count of Units; unit: Hypoglycemic Events
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 16 | 16
Number analyzed (Hypoglycemic Events) | 59 | 56
Hypoglycemic Events | 57 | 54
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.93, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

17. Post Hoc Outcome: Clinical Grading - Initial and 15-min Treatment Correct
Description: as for outcome 16
Time Frame: 60 minutes
Population: Analysis was limited to hypoglycemic events where Initial and 15-min Treatment were correct.
  4 hypoglycemic events were deemed Indeterminate by the graders during the glucagon period.
Measure: Count of Units; unit: Hypoglycemic Events
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 16 | 16
Number analyzed (Hypoglycemic Events) | 69 | 67
Hypoglycemic Events | 66 | 63
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.66, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

18. Post Hoc Outcome: Clinical Grading - Initial Treatment Correct
Description: as for outcome 16
Time Frame: 60 minutes
Population: This analysis included all hypoglycemic events in which the initial treatment and dose were correct, irrespective of the timing of the BG measurements.
  8 hypoglycemic events were deemed Indeterminate by the graders during the glucagon period and 4 during the glucose tabs period.
Measure: Count of Units; unit: Hypoglycemic Events
Units Other Than Participants: Hypoglycemic Events
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
Number analyzed (Participants) | 16 | 16
Number analyzed (Hypoglycemic Events) | 95 | 92
Hypoglycemic Events | 84 | 88
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) vs Glucose Tabs; Test type: Superiority; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 12 weeks.
Groups:
- G-Pen Mini™ (Glucagon Injection): Participants treat non-severe hypoglycemic events with glucagon.
- Glucose Tabs: Participants treat non-severe hypoglycemic events with glucose tabs.
Arm/Group | G-Pen Mini™ (Glucagon Injection) | Glucose Tabs
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Pen Mini™ (Glucagon Injection) (N=20) | Glucose Tabs (N=20)
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Not related to study drug or procedures. Recovered with Sequelae
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Not related to study drug or procedures. Complete Recovery.
Streptococcal Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Not related to study drug or procedures. Occurred during Extension Phase when participant taking both G-Pen Mini and Glucose Tabs. Complete Recovery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No